CLINICAL TRIAL: NCT01504204
Title: Effect of Sample Medication Use and Application Instructions on Adherence to and Efficacy of Treatment of Patients With Mild to Moderate Acne With Epiduo(R) Gel
Brief Title: Effect of Samples on Acne Treatment With Epiduo® Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015374
Record Dates: First submitted 2011-12-28; First posted 2012-01-05 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
Keywords: adherence; adapalene; benzoyl peroxide; sample; topical treatment
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medication with sample and demonstration (Experimental): Subjects will receive a sample tube of the Adapalene + benzoyl peroxide samples with demonstration of how to use it at the first visit.
  Interventions: Drug: Adapalene + benzoyl peroxide samples; Drug: Adapalene + benzoyl peroxide from standard tube
- Medication without samples (Active Comparator): Subjects will receive the Adapalene + benzoyl peroxide from standard tube without a sample or demonstration of proper use of the medication.
  Interventions: Drug: Adapalene + benzoyl peroxide from standard tube

INTERVENTIONS:
Drug: Adapalene + benzoyl peroxide samples — A sample size tube of the study medication, combination adapalene 0.1% plus benzoyl peroxide 2.5% gel, will be provided with instruction on proper application, including demonstration, at the first visit.
  Other Names: Epiduo
  Arms: Medication with sample and demonstration
Drug: Adapalene + benzoyl peroxide from standard tube — Subjects are instructed to apply the combination adapalene 0.1% plus benzoyl peroxide 2.5% gel once daily to all affected areas.
  Other Names: Epiduo

SUMMARY:
The purpose of this study is to compare adherence to treatment and efficacy with Epiduo® Gel in patients with mild to moderate acne who receive a medication sample and instructions on proper application with their stock size medication tube versus patients who receive only the stock size medication tube.

DETAILED DESCRIPTION:
Adapalene Topical Gel is a Vitamin A type product in a water-based gel that is applied to the skin. It is approved by the United States Food and Drug Administration (FDA) for the treatment of acne. Benzoyl Peroxide is a medication applied to the skin that is also approved by the FDA for the treatment of acne and has anti-bacterial properties.

The purpose of this study is to evaluate the safety and effectiveness of a drug called Epiduo® Gel 0.1%/2.5% for the treatment of acne vulgaris.Epiduo® is a combination of adapalene and benzoyl peroxide. This combination drug is approved by the FDA for sale in the United States for use in individuals with acne who are over the age of 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with mild to moderate acne, aged 12 and older, who agrees to participate and provides written consent.
* Have an Acne Global Assessment (AGA) of mild to moderate acne (an AGA score of 2 or 3)

Exclusion Criteria:

* Presence of a concurrent medical condition or skin condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Subjects with known allergy or sensitivity to Epiduo® Gel (or Benzoyl Peroxide Gel) or components therein, including adapalene or benzoyl peroxide
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Reliable methods of birth control are: abstinence (not having sex), oral contraceptives, intrauterine device (IUD), Depo-Provera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Wake Forest Baptist Medical Center Dermatology clinic and phone database of previously seen mild to moderate acne.
Period: Overall Study
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Customized [Median (Full Range); unit: years]
  Age | 19 [13 to 31] | 19 [13 to 29] | 19 [13 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race(Caucasian) | 5 | 6 | 11
  Ethnicity(Non-Hispanic) | 8 | 9 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Study Medication
Description: Adherence will be reported as percentage of prescribed doses taken as measured electronically by a Medication Event Monitoring System (MEMS®) cap.
Time Frame: Baseline to 6 weeks
Population: the median and ranges of subject ages for the sample and no sample group were 19 years, primarily female identifying as Caucasian.
Measure: Median (Standard Deviation); unit: percentage of doses
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples
Number analyzed (Participants) | 9 | 9
percentage of doses | 86 (2.2) | 71 (0.34)

2. Secondary Outcome: Change in Acne Global Assessment
Description: Change in the physician's global assessment of acne severity on a validated 0-5 scale (0=clear to 5=very severe) from baseline to Week 6 visit.
Time Frame: Baseline and 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples
Number analyzed (Participants) | 9 | 9
Participants
  Baseline: AGA (2-mild) | 5 | 6
  Baseline: AGA (3 moderate) | 4 | 3
  Baseline: AGA (1 almost clear) | 0 | 0
  Week 6: AGA (2-mild) | 3 | 4
  Week 6: AGA (3 moderate) | 2 | 3
  Week 6: AGA (1 almost clear) | 4 | 2

3. Secondary Outcome: Change in Acne Lesion Count
Description: Change in total count of acne lesions from baseline visit to Week 6 visit
Time Frame: Baseline and 6 weeks
Measure: Mean (Full Range); unit: lesions
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples
Number analyzed (Participants) | 9 | 9
lesions
  Basleine (Inflammatory Lesions) | 3 [0 to 10] | 2 [0 to 12]
  Baseline (Non-Inflammatory) | 33 [16 to 57] | 38 [6 to 62]
  Week 6 (inflammatory Lesion) | 1 [0 to 9] | 1 [0 to 14]
  Week 6 (Non-inflammatory Lesion) | 19 [5 to 40] | 35 [4 to 53]

ADVERSE EVENTS:
Time Frame: One year
Description: Eighteen subjects completed questionnaires regarding side effects.
Arm/Group | Medication With Sample and Demonstration | Medication Without Samples
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication With Sample and Demonstration (N=10) | Medication Without Samples (N=10)
Dryness (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — Dry skin
itching (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) — Skin itching
redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — red skin

LIMITATIONS AND CAVEATS:
This small pilot study subgroup analyses was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No